CLINICAL TRIAL: NCT05368974
Title: An Observational Study of Mother-Infant Outcomes Following Antenatal Exposure to Direct-Acting Antivirals: the Treatment in Pregnancy for Hepatitis C ("TiP-HepC") Registry
Brief Title: The Treatment in Pregnancy for Hepatitis C ("TiP-HepC") Registry
Acronym: TiP-HepC
Status: Recruiting | Type: Observational
Sponsor: The Task Force for Global Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00083175
Record Dates: First submitted 2022-04-26; First posted 2022-05-10 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis C
Keywords: pregnancy; hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Direct Acting Antivirals — Direct-acting antiviral exposure during documented pregnancy

SUMMARY:
Clinical interventions to reduce the risk of vertical transmission of hepatitis C virus (HCV) infection from mother to infant are highly limited. Direct-acting antiviral (DAA) medications have demonstrated excellent safety and efficacy in non-pregnant individuals, but there is a lack of data regarding the safety of these medications in pregnant women and the effectiveness of these medications in reducing mother-to-child transmission. Therefore, although HCV screening during pregnancy is now recommended in many countries, there is no approved treatment for HCV during pregnancy. An observational study is here proposed to assess outcomes of mother-infant pairs exposed to DAAs during pregnancy within a global clinical case registry. Data regarding the exposures and outcomes of mother-infant pairs exposed to DAAs during pregnancy will be solicited and collected from clinical providers, healthcare facilities, HCV treatment programs, and other clinical practices worldwide. Data will be shared and maintained within a secure database, and cumulative data will be analyzed at pre-determined six-month intervals. The primary outcome will be the number and proportion of mother-infant pairs with adverse pregnancy or birth outcomes. The results of this study will inform HCV treatment decisions by clinical providers and programs worldwide.

DETAILED DESCRIPTION:
In 2016, approximately 6% of all women who were tested for HCV during pregnancy in the United States were HCV antibody-positive. That year, there were 14,417 live births delivered by HCV-positive women, which comprised 0.38% of all live births in the US. Globally, the HCV prevalence among pregnant women varies widely (0.06%-7%) depending on regional and local epidemiology and risk factors. Approximately 5.8% of infants born to HCV-infected mothers will acquire HCV infection with higher rates of transmission among women with HIV co-infection. The primary route for the vertical transmission of HCV is believed to be the perinatal exposure of the infant to maternal blood, though in utero transmission also occurs.

Hepatitis C virus (HCV) testing for pregnant women is now recommended in many countries and universal HCV screening for pregnant women was adopted in the United States in 2020. No clinical interventions have been proven to reduce perinatal HCV transmission, but current and clinical practice guidelines include recommendations for the avoidance of potentially invasive procedures during delivery (ie, chorionic villus sampling, fetal scalp monitoring, episiotomy). The effect of virologic suppression or cure of HCV infection during pregnancy on the risk of mother-to-child HCV transmission has not been directly studied. Previous HCV treatment regimens were contra-indicated in pregnancy due to the inclusion of ribavirin and other teratogenic drugs. More recently, interferon- and ribavirin-free direct-acting antiviral (DAA) medications have raised the potential for HCV treatment during pregnancy to prevent perinatal transmission of HCV and allow for treatment of women during pregnancy. Over half of women reported a preference for HCV treatment during pregnancy if it reduced the probability of vertical transmission to the infant. In addition to potentially reducing vertical transmission to the infant during the current pregnancy, treatment during pregnancy can increase the number of women treated for HCV, and decrease the likelihood of being infected during subsequent pregnancies. Many vulnerable women are at high-risk for loss-to-follow-up following delivery and many women living with HCV may only be eligible for health insurance during pregnancy and immediately postpartum.

Several DAA regimens have demonstrated excellent safety and efficacy profiles in non-pregnant individuals across multiple or all HCV genotypes, achieving cure in >95% of people in as few as 8 weeks of once-daily oral treatment. However, there are limited data regarding the safety and efficacy of DAAs in pregnancy. A phase I pharmacokinetic study of sofosbuvir/ledipasvir (SOF/LDV) in 9 pregnant women demonstrated similar drug levels to non-pregnant individuals with excellent safety and efficacy profile, and a similar study of sofosbuvir/velpatasvir (SOF/VEL) is currently enrolling participants. A prospective study of 15 women treated with SOF/LDV in India reported no adverse events. No other trials have been conducted or registered for pregnant individuals to date. The frequency and outcomes for women who become pregnant while on DAA treatment have been rarely reported. Currently, there is only one published study reporting outcomes of mother-infant pairs of women who became pregnant while on DAA treatment; among 100 women, 9 of whom completed 12 weeks of treatment with various regimens, no major adverse events were reported.

Given the paucity of data regarding the safety and efficacy of DAA treatment in pregnancy, the American College of Obstetrics and Gynecology and Society for Maternal-Fetal Medicine recommend that DAAs "only be initiated in the setting of a clinical trial during pregnancy and that people who become pregnant while taking a direct-acting antiviral should be counseled in a shared decision-making framework about the risks and benefits of continuation." The Infectious Diseases Society of America and the American Association for the Study of Liver Diseases (IDSA/AASLD) advise that "treatment can be considered during pregnancy on an individual basis after a patient-physician discussion about the potential risks and benefits". Treatment for HCV in pregnancy therefore remains an off-label use of DAA medications and clinical practices remain highly variable by providers and programs. The frequency, geographic distribution, safety profile or effectiveness of HCV treatment during pregnancy for mother-infant pairs have not been evaluated or reported.

The primary objective of this observational study is to assess the safety of DAA treatment in mother-infant pairs with exposure to DAA medications during pregnancy within a clinical case registry. The secondary objectives of this study are to describe the frequency and distribution of known cases of DAA exposure during pregnancy and to assess the effectiveness of DAA treatment in pregnancy in achieving HCV cure for mothers and reducing the transmission of HCV from mother to infant.

This is an observational study of the outcomes of mother-infant pairs exposed to DAA treatment during pregnancy in routine clinical practice using de-identified data from a convenience sample of health facilities, public health, government, and private entities globally. Data regarding the demographics, baseline clinical status, timing and type of DAA exposure, and pregnancy/birth outcomes of mother-infant pairs exposed to DAAs during pregnancy will be solicited from clinical providers, health facilities, HCV treatment programs, and other clinical practices or programs prescribing DAA treatment. Data will be coded, standardized, and pooled in a common database for analysis.

ELIGIBILITY:
Inclusion Criteria:

-Documented pregnancy with: Estimated date of conception by documentation of either 1) date of last menstrual period or 2) ultrasound evaluation Actual date of delivery

* Documented chronic HCV infection prior to or during pregnancy (positive test for HCV RNA or HCV core antigen)
* Documented DAA exposure occurring within 30 days of the estimated date of conception and before the pregnancy outcome (ie, fetal demise, spontaneous abortion, live delivery, etc). Eligible DAA drugs are listed in Appendix 1.

Exclusion Criteria:

- DAA exposures that include ribavirin or interferon will be excluded given their established harm during pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with chronic HCV infection and documented pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse pregnancy outcomes | 1 year
  The primary outcomes measured in the study are adverse pregnancy and birth outcomes documented at the time of the outcome of the pregnancy (primary endpoint). Primary adverse pregnancy outcomes include preterm delivery (<37 weeks gestational age), stillbirth or fetal demise, and maternal death.
Number of adverse birth outcomes | 1 year
  Primary adverse birth outcomes include low birth weight (<2500g), small for gestational age, need for neonatal intensive care, and presence of congenital anomaly.

SECONDARY OUTCOMES:
Proportion of registry participants achieving SVR12 | 12 weeks
  Secondary outcomes of the study are the proportion of women achieving HCV cure by HCV PCR test 12 weeks following last DAA treatment (SVR12)
Proportion of infants with HCV infection | 18 months
  proportion of infants with evidence of chronic HCV infection after 2 months of age by HCV PCR or after 18 months of age by anti-HCV antibody seropositivity

CONTACTS AND LOCATIONS:
Overall Officials: John Ward, MD, Principal Investigator — The Taskforce For Global Health
Locations (1):
- The Taskforce for Global Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AASLD & IDSA. HCV Guidance: Recommendations for Testing, Managing, and Treating Hepatitis C, v2021.1.
- [Background] AbdAllah M, Alboraie M, Abdel-Razek W, Hassany M, Ammar I, Kamal E, Alalfy M, Okasha A, El Akel W, Shaaban E, Elbaz T, Hefny Z, Gomaa A, El-Bendary M, El-Serafy M, Esmat G, Doss W, El-Sayed MH. Pregnancy outcome of anti-HCV direct-acting antivirals: Real-life data from an Egyptian cohort. Liver Int. 2021 Jul;41(7):1494-1497. doi: 10.1111/liv.14913. Epub 2021 May 11. PMID 33905164
- [Background] Benova L, Mohamoud YA, Calvert C, Abu-Raddad LJ. Vertical transmission of hepatitis C virus: systematic review and meta-analysis. Clin Infect Dis. 2014 Sep 15;59(6):765-73. doi: 10.1093/cid/ciu447. Epub 2014 Jun 13. PMID 24928290
- [Background] Chappell CA, Scarsi KK, Kirby BJ, Suri V, Gaggar A, Bogen DL, Macio IS, Meyn LA, Bunge KE, Krans EE, Hillier SL. Ledipasvir plus sofosbuvir in pregnant women with hepatitis C virus infection: a phase 1 pharmacokinetic study. Lancet Microbe. 2020 Sep;1(5):e200-e208. doi: 10.1016/S2666-5247(20)30062-8. Epub 2020 Jul 27. PMID 32939459
- [Background] Cottrell EB, Chou R, Wasson N, Rahman B, Guise JM. Reducing risk for mother-to-infant transmission of hepatitis C virus: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 Jan 15;158(2):109-13. doi: 10.7326/0003-4819-158-2-201301150-00575. PMID 23437438
- [Background] Kushner T, Cohen J, Tien PC, Terrault NA. Evaluating Women's Preferences for Hepatitis C Treatment During Pregnancy. Hepatol Commun. 2018 Oct 1;2(11):1306-1310. doi: 10.1002/hep4.1264. eCollection 2018 Nov. PMID 30411077
- [Background] Kushner T, Reau N. Changing epidemiology, implications, and recommendations for hepatitis C in women of childbearing age and during pregnancy. J Hepatol. 2021 Mar;74(3):734-741. doi: 10.1016/j.jhep.2020.11.027. Epub 2020 Nov 25. PMID 33248169
- [Background] Mok J, Pembrey L, Tovo PA, Newell ML; European Paediatric Hepatitis C Virus Network. When does mother to child transmission of hepatitis C virus occur? Arch Dis Child Fetal Neonatal Ed. 2005 Mar;90(2):F156-60. doi: 10.1136/adc.2004.059436. PMID 15724041
- [Background] Schillie SF, Canary L, Koneru A, Nelson NP, Tanico W, Kaufman HW, Hariri S, Vellozzi CJ. Hepatitis C Virus in Women of Childbearing Age, Pregnant Women, and Children. Am J Prev Med. 2018 Nov;55(5):633-641. doi: 10.1016/j.amepre.2018.05.029. PMID 30342628
- [Background] Schillie S, Wester C, Osborne M, Wesolowski L, Ryerson AB. CDC Recommendations for Hepatitis C Screening Among Adults - United States, 2020. MMWR Recomm Rep. 2020 Apr 10;69(2):1-17. doi: 10.15585/mmwr.rr6902a1. PMID 32271723
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Dotters-Katz SK, Kuller JA, Hughes BL. Society for Maternal-Fetal Medicine Consult Series #56: Hepatitis C in pregnancy-updated guidelines: Replaces Consult Number 43, November 2017. Am J Obstet Gynecol. 2021 Sep;225(3):B8-B18. doi: 10.1016/j.ajog.2021.06.008. Epub 2021 Jun 8. PMID 34116035
- [Background] Yattoo G. Treatment of chronic hepatitis C with ledipasvir/sofosbuvir combination during pregnancy. Hepatol Int. 2018;12(Suppl. 2):S292-3.